CLINICAL TRIAL: NCT02242929
Title: Surgical Excision Versus Combined Treatment With Curettage and Imiquimod for Nodular Basal Cell Carcinoma: an Open, Non-inferiority, Randomized Controlled Trial
Brief Title: Surgery Versus Combined Treatment With Curettage and Imiquimod for Nodular Basal Cell Carcinoma
Acronym: SCIN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL50433.068.14
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Nodular Basal Cell Carcinoma
Keywords: Nodular Basal Cell Carcinoma; Treatment; Imiquimod; Curettage; Surgery
MeSH Terms: interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard surgical excision (Active Comparator): Standard surgical "elliptical" excision including a 3-mm clinically tumour-free margin according to the current local hospital arrangements.
  Interventions: Procedure: Standard surgical excision
- Imiquimod 5% cream with prior curettage (Experimental): Tumours will be partially debulked under local anaesthesia by removing all tumour tissue until normal dermis remains with a blunt curette. After curettage patients will receive an instruction sheet to apply imiquimod 5% cream once daily, 5 days a week, during 6 weeks, starting one week after the curettage procedure. Patients will be instructed to apply a thin layer to the tumour including 5-10mm of the surrounding skin at least 1 hour before going to bed at night. The lesion will not be covered (unless needed because of weeping or bleeding). Participants will be asked to wash their hands after applying the cream, and to wipe the cream off after 8 hours (in the morning).
  Interventions: Drug: Imiquimod 5% cream with prior curettage

INTERVENTIONS:
Drug: Imiquimod 5% cream with prior curettage
  Other Names: Aldara
  Arms: Imiquimod 5% cream with prior curettage
Procedure: Standard surgical excision
  Arms: Standard surgical excision

SUMMARY:
Basal cell carcinoma (BCC) is a slow-growing, locally invasive malignant epidermal skin tumour. It is the most common malignant disease in Caucasians, representing approximately 80% of all cases of skin cancer and is therefore an important health problem. In the Netherlands incidence rates are 165 for men and 157 for women per 100.000 person-years, and these rates are rising with 3-10% every year.

A simplified histological classification of BCCs includes the following three subtypes: nodular, superficial and infiltrative variants, with the nodular variant being the most frequent type. Although a characteristic feature of BCCs is their low risk to metastasize, if untreated they may be locally invasive and may induce considerable functional and cosmetic morbidity.

The gold standard treatment of all histological BCC subtypes is surgical excision (SE), but not all patients are eligible for surgery. In patients with multiple BCCs and older patients, surgery may lead to significant morbidity, and in some cases, it may result in disfiguring scarring. For these reasons and to reduce workload and costs in the healthcare system, there is a growing demand for alternative, non-invasive, treatments. An advantage of non-invasive treatment options is that they can be performed by other healthcare professionals, such as general practitioners and specialized nurses. For treatment of superficial BCCs (sBCC) non-invasive treatments, such as topical imiquimod (IMQ), 5-fluorouracil (5-FU) or photodynamic therapy (PDT) are already commonly used. Our group investigated the efficacy of those three therapies and found that after 3 years, BCCs treated with IMQ had a significant lower risk of recurrence, compared to the other therapies.

A recent study suggests that IMQ, besides being an immune-response modifier, also directly inhibits sonic hedgehog (SHH) signalling, the most important pathway active in BCCs. This targeted effect of IMQ very likely explains the superior therapeutic effect. Treatment of nodular BCC (nBCC) with IMQ has been investigated. Without prior curettage, high efficacy rates were found, although efficacy was still slightly inferior to SE.

The investigators hypothesize that the effectiveness of IMQ following prior curettage will not be inferior to SE and that the benefits will be a higher patient satisfaction and lower healthcare costs. A recently published discreet choice experiment showed that patients preferred IMQ to surgery regardless of previous experience of BCC symptoms and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Primary histologically proven nodular BCC ≥ 4mm and ≤ 20mm in diameter. (If the tumour exhibits additional sBCC characteristics, but also contains nodular component that extend into the reticular dermis, the tumour will be classified as nBCC with superficial components and will be included).
* Comorbidities may not interfere with study treatment
* Capable to understand instructions

Exclusion Criteria:

* A nodular BCC located in the H-zone of the face or hairy scalp
* Recurrent (previously treated) nBCC
* Aggressive BCC subtypes (morphoea, micronodular, or BCC with squamous differentiation)
* Life expectancy of less than five years
* Breast-feeding or pregnant women
* Serious comorbidities
* Use of immunosuppressive medication during the trial period or within 30 days before enrolment
* Patients with genetic skin cancer disorders

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants tumour-free | At 1 year after end of treatment
  The primary study endpoint is the proportion of participants tumour-free at 1 year after end of treatment (defined as absence of initial treatment failure or any clinical signs of local recurrence). For SE, routine histological examination of haematoxylin and eosin (H&E)-stained sections of the lateral and deep margins will be used to assess treatment failure. For curettage & IMQ 5% cream, initial treatment failure will be clinically assessed at a follow-up visit 3 months after end of treatment. Initial treatment failure or any clinical signs of subsequent local recurrence will be assessed and recorded separately by one investigator. In case there is clinical suspicion of BCC, a 3 mm punch biopsy will be taken for histological verification.

SECONDARY OUTCOMES:
The 5-year cumulative probability of recurrence free survival after end of treatment | At 5 years after end of treatment
  Any clinical signs of subsequent local recurrence will be assessed by one investigator. In case there is clinical suspicion of BCC, a 3 mm punch biopsy will be taken for histological verification.
Compliance | At 3 months after end of treatment
  Data for compliance with the prescribed regimens of IMQ 5% cream will be obtained from a personal diary kept by patients and completed daily during the six week IMQ 5% application period in subjects allocated to treatment with IMQ. Compliance will be calculated as the number of applications actually applied by the patient divided by the total prescribed number of cream applications. Furthermore sachets will be collected and counted by the investigator. This is a separate compliance assessment. The number of returned sachets will be divided by the total prescribed number of sachets. During the phone consultation by the investigator two weeks after start of application, treatment will be evaluated to ensure continuation of treatment.
Cosmetic appearance | At 1 and 5 year after end of treatment
  Cosmetic appearance of lesion site will be assessed independently by the participant and two independent investigators at 1 and 5 year follow-up using a Dutch four point scale and the Patient and Observer Scar Assessment Scale (POSAS).
Patient satisfaction | At 1 and 5 year after end of treatment
  Patient satisfaction will be assessed by the participant at 1 and 5 year follow-up on the basis of 3 statements. For the extent of agreement a 4-point rating scale is used, ranging from total disagreement to total agreement
Level of Pain | 2 weeks after end of treatment
  The proportion of patients experiencing a moderate or more severe level of pain. In the IMQ 5 % group, this will be measured daily during the application period and 2 weeks after end of treatment. In the SE group, pain during SE procedure will be measured and pain until the removal of the stiches will be measured daily. Furthermore pain will be measured at the time of removal of the stiches. Pain will be assessed using a 10 cm Visual Analogue Scale (VAS) where 0 represents 'no pain' and 10 represents, 'most severe pain imaginable'.
Cost-effectiveness | At 5 year after end of treatment
  Data regarding resource use, i.e. outpatient visits, phone consultation, curettage, IMQ cream, SE and potential treatment of side-effects/adverse events will be recorded during the trial. Cost-prices will be derived from the manual for cost research in economic evaluations, the Pharmacotherapeutic Compass and the university hospital Maastricht. If necessary, cost-prices will be calculated based on real resource use. Total treatment costs will be estimated by multiplying volumes of use with the costs per unit. The cost-effectiveness ratio will be expressed as the incremental costs per additional tumour free patient. To quantify the uncertainty surrounding the incremental cost-effectiveness ratio (ICER) bootstrap analysis will be performed. Results of this analysis will be presented in cost-effectiveness planes and acceptability curves.
Adverse events | Up to 3 months after end of treatment
  Adverse events, including local skin reactions, will be collected from all patients up to the 3 months follow-up visit and during phone consultation by the investigator (after two weeks of treatment in the IMQ group and during phone consultation about the histological examination of the excision specimen in the SE group). In case of an extra (phone) consultation of the patients as a result of severe adverse reactions, this will also be recorded. Serious events related to the investigative treatments (SUSAR) will be recorded during the entire follow-up period.

OTHER OUTCOMES:
Baseline characteristics | After inclusion visit
  Baseline characteristics (ie. age, sex, amount of sun-exposure, size and localisation of the target tumour, medical history and concomitant medication) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Mosterd, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Bath-Hextall F, Ozolins M, Armstrong SJ, Colver GB, Perkins W, Miller PS, Williams HC; Surgery versus Imiquimod for Nodular Superficial basal cell carcinoma (SINS) study group. Surgical excision versus imiquimod 5% cream for nodular and superficial basal-cell carcinoma (SINS): a multicentre, non-inferiority, randomised controlled trial. Lancet Oncol. 2014 Jan;15(1):96-105. doi: 10.1016/S1470-2045(13)70530-8. Epub 2013 Dec 11. PMID 24332516
- [Derived] Verkouteren BJA, Nelemans PJ, Sinx KAE, Kelleners-Smeets NWJ, Winnepenninckx VJL, Arits AHMM, Mosterd K. Imiquimod Cream Preceded by Superficial Curettage vs Surgical Excision for Nodular Basal Cell Carcinoma: A Secondary Analysis of a Randomized Clinical Trial. JAMA Dermatol. 2025 Mar 1;161(3):299-304. doi: 10.1001/jamadermatol.2024.5572. PMID 39878970
- [Derived] Sinx KAE, Nelemans PJ, Kelleners-Smeets NWJ, Winnepenninckx VJL, Arits AHMM, Mosterd K. Surgery versus combined treatment with curettage and imiquimod for nodular basal cell carcinoma: One-year results of a noninferiority, randomized, controlled trial. J Am Acad Dermatol. 2020 Aug;83(2):469-476. doi: 10.1016/j.jaad.2020.04.053. Epub 2020 Apr 19. PMID 32320773